CLINICAL TRIAL: NCT04858451
Title: Community Participants With COPD or Bronchiectasis and at Risk of Respiratory Viral Infections Including SARS-CoV-2: An Open-label, Multicentre Feasibility Study of an Inhaled Nitric Oxide Generating Solution (RESP301)
Brief Title: COmmunity Patients at Risk of Viral Infections Including SARS-CoV-2
Acronym: CORVIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopping criteria were met. A safety event has occurred which was classified as an SAE and was related to the study intervention.
Sponsor: Thirty Respiratory Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RESP301-005
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: COPD; Bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Part 1a: Dose Finding Phase
  Up to 48 eligible participants will be administered single ascending doses of RESP301 to determine the maximum tolerated dose, according to the following schedule:
  * 8 participants to receive RESP301 at a dose of 1 ml
  * 8 participants to receive RESP301 at a dose of 2 ml
  * 8 participants to receive RESP301 at a dose of 3 ml
  * 8 participants to receive RESP301 at a dose of 4 ml
  * 8 participants to receive RESP301 at a dose of 5 ml
  * 8 participants to receive RESP301 at a dose of 6 ml
  Part 1b: Concomitant Medication Expansion Phase
  • 8 participants to receive RESP301 at MTD with short-acting bronchodilator administered 10min prior to RESP301
  Part 2: Expansion Phase
  A minimum of 150 patients will be enrolled in to the Expansion Phase. These may include eligible participants from Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): In Part 1a, up to 48 patients will be administered single ascending doses of RESP301 (1-6ml; 8 patients per dose cohort). Provided that individual stopping criteria are not met in ≥3 participants, and there are no serious adverse events that are at least possibly related to RESP301, the next dose cohort can be enrolled. Patients can be enrolled into more than one dose cohort provided they did not meet individual stopping criteria.
  In Part 1b, 8 participants will receive RESP301 at MTD determined in Part 1a, with short-acting bronchodilator administered 10min prior to RESP301.
  In Part 2, a minimum of 150 patients will be enrolled. This may include patients who took part in Part 1. At least the first 50 patients will receive a test dose of RESP301 before enrolment into the "dormant phase". Patients who experience flare-up symptoms while in the dormant phase, may proceed to the treatment phase where they will self-administer RESP301 at home for 7 days.
  Interventions: Drug: RESP301

INTERVENTIONS:
Drug: RESP301 — A single RESP301 dose administered at a study site to assess tolerability.
  In patients who experience a flare-up during the study period, self-administered RESP301 treatment for 7 days, 3 times a day.

SUMMARY:
Patients with a respiratory disease are at higher risk of poor outcomes due to worsening of symptoms caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) and other respiratory infections. New therapies are needed for treating high risk patients at early stages of an infection. This study will assess the safety, tolerability and feasibility of using an inhaled nitric oxide generating solution, RESP301, as a self-administered treatment following flare-up of symptoms.

RESP301 is a liquid solution which produces nitric oxide in the lungs when inhaled using a nebuliser. The components of RESP301 are already used in clinical practice and inhaled nitric oxide is used as a treatment for newborns and patients with Chronic Obstructive Pulmonary Disease (COPD). In a laboratory setting, RESP301 has been shown to be effective against respiratory viruses, including SARS-CoV-2.

This study will first determine the maximum tolerated dose of RESP301 in up to 48 adult patients with COPD or bronchiectasis in the United Kingdom (UK) (Part 1a; Dose Finding Phase). Once the Maximum Tolerated Dose (MTD) has been determined in Part 1a, a cohort of 8 patients will be recruited and RESP301 administered at the MTD but these patients will in addition receive a single dose of a short acting bronchodilator 10 minutes preceding administration of RESP301.

After completion of Part 1, approximately 150 patients will be recruited into Part 2 of the trial (Expansion Phase). A minimum of 50 participants will receive a test dose of RESP301 during a screening visit. Response to the test dose will be monitored. Participants who tolerate the test dose will continue in the study and should contact the study team if they experience exacerbation symptoms in the next 52 weeks. Following a call with the site team to discuss symptoms, participants will receive RESP301 delivered to their home to self-administer for 7 days. The study duration for each participant will be at most 57 weeks, including the study visit and monthly calls. Participants who start the course of study treatment, will receive daily calls during the treatment period and will also be followed up after they complete the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female of non-childbearing potential or male ≥35 years of age, at the time of signing the informed consent
2. Able and willing to provide informed consent
3. Spirometry-confirmed diagnosis of COPD (FEV1/FVC<0.7 post-bronchodilator) or computerised tomography (CT) proven bronchiectasis
4. Part 1 only: FEV1 ≥50% predicted at screen 1 (i.e. FEV1 prior to any in-clinic administered short acting bronchodilator)

Exclusion Criteria:

1. Unable to safely use a nebuliser as required by the study according to Investigator's opinion
2. Severe COPD or bronchiectasis defined as FEV1 <20% or requiring non-invasive ventilation
3. History of methaemoglobinaemia
4. Baseline methaemoglobin concentration (using fingertip sensor) > 2%
5. Uncontrolled or severe asthma or history of severe bronchospasm
6. Presence of tracheostomy/inability to provide spirometry or contraindication for performing spirometry
7. Allergy to any of the components of the study intervention
8. Participation in other clinical investigations utilising investigational treatment within the last 30 days / 5 half lives whichever is longer
9. Deemed unlikely to be able to adhere to protocol in view of investigator
10. Any subject who in the opinion of the investigator would not be best served by participating in this clinical trial
11. Any unstable, uncontrolled or severe medical condition which in the opinion of the investigator would make the patient unsuitable for the trial
12. Participant lives at home with no other adults in the household (Part 2 only)
13. On long-term non-invasive ventilation and/or at higher risk of bronchospasm
14. Prescribed Nitric Oxide donating agent (Nitroprusside, Isosorbide dinitrate, Isosorbide mononitrate, Naproxcinod, Molsidomine and Linsidomine)
15. Female of childbearing potential
16. Clinical diagnosis of COPD but Screening Visit spirometry at study centre excludes COPD (i.e. FEV1/FVC post bronchodilator ratio is not <0.7)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Medicines Evaluation Unit, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: total 13 participants enrolled in Part 1A and 10 participants were enrolled in more than one cohort
Groups:
- Part 0: Based on Protocol Version 3.0
- Part 1A - SAD 1ml: Participants were administered single dose of 1ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - SAD 2ml: Participants were administered single dose of 2ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - SAD 3ml: Participants were administered single dose of 3ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - SAD 4ml: Participants were administered single dose of 4ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - SAD 5ml: Participants were administered single dose of 5ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - SAD 6ml: Participants were administered single dose of 6ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1B - MTD 6ml: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD determined in Part 1a) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 2 - RTD 4ml: Participants were administered a single test dose of RESP301 at the RTD of 4 mL. if tolerated and symptoms of exacerbation developed, eligible participants were to self-administer RESP301 TID for 7 days at the RTD.
Period: Part 0 (Protocol Version 3.0)
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 1ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 2ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 3ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 4ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 5ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A - 6ml
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1B
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 0 | Part 1A - SAD 1ml | Part 1A - SAD 2ml | Part 1A - SAD 3ml | Part 1A - SAD 4ml | Part 1A - SAD 5ml | Part 1A - SAD 6ml | Part 1B - MTD 6ml | Part 2 - RTD 4ml
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
Not completed — Discontinued | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63

BASELINE CHARACTERISTICS:
Population: participants who received at least one dose of RESP301.
Groups:
- Part 0: Patients who were enrolled under protocol version 3.0
- Part 1A: Participants were administered single ascending dose of RESP301 from 1ml to 6ml in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1B: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 2: Participants were administered a single test dose of RESP301 at the RTD of 4 mL. if tolerated and symptoms of exacerbation developed, eligible participants were to self-administer RESP301 TID for 7 days at the RTD.
- Total: Total of all reporting groups
Arm/Group | Part 0 | Part 1A | Part 1B | Part 2 | Total
Number analyzed (Participants) | 4 | 13 | 8 | 16 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (5.07) | 68.2 (6.11) | 67.6 (4.78) | 65.3 (9.13) | 66.9 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 4 | 10 | 23
  Male | 2 | 6 | 4 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 13 | 8 | 16 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 2 | 3 | 2 | 3 | 10
  Former smoker | 2 | 10 | 6 | 11 | 29
  Never smoked | 0 | 0 | 0 | 2 | 2
Height [Mean (Standard Deviation); unit: m] | 1.663 (0.0608) | 1.648 (0.1049) | 1.664 (0.1119) | 1.664 (0.1007) | 1.659 (0.0981)
Weight [Mean (Standard Deviation); unit: kg] | 89.53 (20.128) | 75.90 (10.992) | 85.19 (14.750) | 83.31 (19.178) | 81.93 (16.207)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 32.650 (8.6157) | 27.954 (3.5671) | 30.600 (2.8894) | 30.144 (7.3258) | 29.783 (5.7503)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Tolerating RESP301 at Each Dose Level in Part 1
Description: Defined as percentage of participants able to tolerate the test dose, i.e. able to complete the test dose without any of the following:
  * Troublesome cough, chest pain or tightness, bronchospasm or dyspnoea that is deemed unacceptable by the patient
  * methaemoglobin >5% during or >3% post dose (60 mins)
  * any treatment-related AE that led to participant not being able to complete the test dose
  * >20% reduction in FEV1 pre dose to post dose at 60min if additionally reporting troublesome cough, chest pain or tightness, bronchospasm or dyspnoea that is deemed unacceptable by the patient
Time Frame: Screening Visit
Population: participants who received at least one dose of RESP301
Measure: Count of Participants; unit: Participants
Groups:
- SAD-1ml: Participants were administered single dose of 1ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 2ml: Participants were administered single dose of 2ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 3ml: Participants were administered single dose of 3ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 4ml: Participants were administered single dose of 4ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 5ml: Participants were administered single dose of 5ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 6ml: Participants were administered single dose of 6ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- MTD 6ml +SABA MTD 6ml +SABA MTD 6ml +SABA: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
Arm/Group | SAD-1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml +SABA MTD 6ml +SABA MTD 6ml +SABA
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8
Participants | 8 | 8 | 8 | 8 | 8 | 6 | 8

2. Primary Outcome: Feasibility of Self-administering RESP301 Treatment in Terms of Commencing Treatment
Description: Defined as percentage of patients who, having experienced and correctly reported an exacerbation, commence self-administration of the treatment on the day the treatment is delivered
Time Frame: 1 day
Population: Due to early termination of the study, no participants entered the Treatment Period of Part 2, and therefore no feasibility of self administering RESP301 data was collected.
Groups:
- All Participants: In Part 1a, up to 48 patients will be administered single ascending doses of RESP301 (1-6ml; 8 patients per dose cohort). Provided that individual stopping criteria are not met in ≥3 participants, and there are no serious adverse events that are at least possibly related to RESP301, the next dose cohort can be enrolled. Patients can be enrolled into more than one dose cohort provided they did not meet individual stopping criteria.
  In Part 1b, 8 participants will receive RESP301 at MTD determined in Part 1a, with short-acting bronchodilator administered 10min prior to RESP301.
  In Part 2, a minimum of 150 patients will be enrolled. This may include patients who took part in Part 1. At least the first 50 patients will receive a test dose of RESP301 before enrolment into the "dormant phase". Patients who experience flare-up symptoms while in the dormant phase, may proceed to the treatment phase where they will self-administer RESP301 at home for 7 days.
  RESP301: A single RESP301 dose administered at a study site to assess tolerability.
  In patients who experience a flare-up during the study period, self-administered RESP301 treatment for 7 days, 3 times a day.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Primary Outcome: Feasibility of Self-administering RESP301 Treatment in Terms of Treatment Compliance
Description: For those participants commencing self-administration of RESP301, the percentage of total doses taken
Time Frame: 7 days
Population: as for outcome 2
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Tolerability of RESP301 (in Part 1a, Part 1b, and Part 2)
Description: Defined as percentage of participants able to tolerate the test dose, i.e. able to complete the test dose without any of the following:
  * Troublesome cough, chest pain or tightness, bronchospasm or dyspnoea that is deemed unacceptable by the patient
  * methaemoglobin >5% during or >3% post dose (60 mins)
  * any treatment-related AE that led to participant not being able to complete the test dose, and/or be suitable to be enrolled into the dormant phase in the Investigator's opinion
  * for the first 50 patients who will undergo pre spirometry, >20% reduction in FEV1 from pre test dose to post test dose with symptoms (patients with >20% reduction in FEV1 without symptoms would be offered the option to continue in the study)
Time Frame: Screening Visit
Population: participants who received at least one dose of RESP301.
Measure: Count of Participants; unit: Participants
Groups:
- SAD - 1ml: Participants were administered single dose of 1ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- RTD - 4ml: Participants were administered a single test dose of RESP301 at the RTD of 4 mL. if tolerated and symptoms of exacerbation developed, eligible participants were to self-administer RESP301 TID for 7 days at the RTD.
Arm/Group | SAD - 1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml +SABA MTD 6ml +SABA MTD 6ml +SABA | RTD - 4ml
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Participants | 8 | 8 | 8 | 8 | 8 | 4 | 7 | 12

5. Secondary Outcome: Safety of RESP301 in Terms of Treatment Emergent Adverse Events
Description: Defined as total counts and cumulative incidence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Parts 1A/1B: Screening/dosing period 1-2 days + Follow-up period 1 day. Part 2: Screening period 1-2days (Participants did not enter the treatment phase due to early study termination)
Population: all participants who consented to the study
Measure: Number; unit: # Events
Groups:
- SAD - 1ml: Participants will be administered single dose of 1ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 2ml: Participants will be administered single dose of 2ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 3ml: Participants will be administered single dose of 3ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 4ml: Participants will be administered single dose of 4ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 5ml: Participants will be administered single dose of 5ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- SAD - 6ml: Participants will be administered single dose of 6ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- MTD 6ml +SABA: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- RTD 4ml: Participants were administered a single test dose of RESP301 at the RTD of 4 mL. if tolerated and symptoms of exacerbation developed, eligible participants were to self-administer RESP301 TID for 7 days at the RTD.
Arm/Group | SAD - 1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml +SABA | RTD 4ml
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 63
# Events | 4 | 7 | 3 | 8 | 10 | 13 | 13 | 16

6. Secondary Outcome: Safety of RESP301 in Terms of Serious Adverse Events
Description: Defined as total counts and cumulative incidence of Serious Adverse Events (SAEs)
Time Frame: as for outcome 5
Population: all participants who consented to the study
Measure: Number; unit: # Events
Arm/Group | SAD - 1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml +SABA | RTD - 4ml
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 63
# Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

7. Secondary Outcome: Safety of RESP301 in Terms of Suspected Unexpected Serious Adverse Reactions
Description: Defined as total counts and cumulative incidence of Suspected Unexpected Serious Adverse Reactions (SUSARs)
Time Frame: as for outcome 5
Population: participants who received at least one dose of RESP301.
Measure: Number; unit: # Events
Groups:
- MTD 6ml + SABA: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
Arm/Group | SAD - 1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml + SABA | RTD 4ml
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
# Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Safety of RESP301 in Terms of Treatment-related AEs
Description: Defined as total counts and cumulative incidence of treatment-related AEs
Time Frame: as for outcome 5
Population: participants who received at least one dose of RESP301.
Measure: Number; unit: # Events
Groups:
- SAD - 5ml; SAD - 6ml: Participants were administered single dose of 6ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
Arm/Group | SAD - 1ml | SAD - 2ml | SAD - 3ml | SAD - 4ml | SAD - 5ml | SAD - 6ml | MTD 6ml +SABA | RTD 4ml
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
# Events | 4 | 4 | 2 | 7 | 8 | 12 | 12 | 16

9. Secondary Outcome: Efficacy of RESP301 in Terms of Percentage of Patients Recovered by Day 7
Description: Defined as percentage of participants recovered by Day 7 post starting treatment, where recovery is defined as patient feels all their symptoms are back to their usual baseline (all symptom Visual Analogue Scores are 0 on a scale from 0 to 10, where 0 is "same as usual" and 10 is "much more than usual")
Time Frame: 7 days
Population: Due to early termination of the study, no participants entered the Treatment Period of Part 2, and therefore no efficacy data was collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Efficacy of RESP301 in Terms of Percentage of Patients Recovered by Day 14
Description: Defined as percentage of participants recovered by Day 14 post starting treatment, where recovery is defined as patient feels all their symptoms are back to their usual baseline (all symptom Visual Analogue Scores are 0 on a scale from 0 to 10, where 0 is "same as usual" and 10 is "much more than usual")
Time Frame: 7 days
Population: Due to early termination of the study, data were not collected and efficacy could not be analysed
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Efficacy of RESP301 in Terms of Time to Recovery
Description: Defined as days to recovery, where recovery is defined as patient feels all their symptoms are back to their usual baseline (all symptom Visual Analogue Scores are 0 on a scale from 0 to 10, where 0 is "same as usual" and 10 is "much more than Defined as percentage of participants recovered by Day 14 post starting treatment, where recovery is defined as patient feels all their symptoms are back to their usual baseline (all symptom Visual Analogue Scores are 0 on a scale from 0 to 10, where 0 is "same as usual" and 10 is "much more than usual")
Time Frame: 21 days
Population: as for outcome 9
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Efficacy of RESP301 in Terms of Preventing Exacerbation-related Hospitalisation and/or Death
Description: Number of patients treated with RESP301 that experience exacerbation-related hospitalisation and/or death
Time Frame: 7 days
Population: as for outcome 9
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Efficacy of RESP301 in Terms of Patient-reported Symptoms
Description: Change in Clinical COPD Questionnaire (CCQ) score from Day 1 to Day 7, where the minimum score is 0 (very good health status) and maximum score is 6 (extremely poor health status)
Time Frame: 7 days
Population: as for outcome 9
Arm/Group | All Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Feasibility of Self-administering RESP301 Treatment in Terms of Receiving Treatment
Description: Defined as percentage of patients who, having experienced and correctly reported an exacerbation, receive the treatment within 48 hours of reporting their exacerbation
Time Frame: 2 days
Population: as for outcome 2
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Part 0: Screening/baseline visit Day 0. Parts 1A/1B: Screening/dosing period 1-2 days + Follow-up period 1 day. Part 2: Screening period 1-2days (Participants did not enter the treatment phase due to early study termination)
Groups:
- Part 1A - 1ml: In Part 1a, up to 48 patients will be administered single ascending doses of RESP301 (1-6ml; 8 patients per dose cohort). Provided that individual stopping criteria are not met in ≥3 participants, and there are no serious adverse events that are at least possibly related to RESP301, the next dose cohort can be enrolled. Patients can be enrolled into more than one dose cohort provided they did not meet individual stopping criteria.
  In Part 1b, 8 participants will receive RESP301 at MTD determined in Part 1a, with short-acting bronchodilator administered 10min prior to RESP301.
  In Part 2, a minimum of 150 patients will be enrolled. This may include patients who took part in Part 1. At least the first 50 patients will receive a test dose of RESP301 before enrolment into the "dormant phase". Patients who experience flare-up symptoms while in the dormant phase, may proceed to the treatment phase where they will self-administer RESP301 at home for 7 days.
  RESP301: A single RESP301 dose administered at a study site to assess tolerability.
  In patients who experience a flare-up during the study period, self-administered RESP301 treatment for 7 days, 3 times a day.
- Part 1A - 2ml: Participants were administered single dose of 2ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - 3ml: Participants were administered single dose of 3ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - 4ml: Participants were administered single dose of 4ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - 5ml: Participants were administered single dose of 5ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 1A - 6ml: Participants were administered single dose of 6ml RESP301 in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events
- Part 1B - 6ml +SABA: Participants were administered short-acting inhaled bronchodilator (2 inhalations of Ventolin - 100mcg per inhalation) through a spacer device 10 minutes before receiving RESP301 and a single dose of 6ml RESP301 (MTD) in the clinic on Day 1, with a follow up safety phone call being conducted on the morning of Day 2 to check for any adverse events.
- Part 2 - RTD 4ml RTD 4ml RTD 4ml: Participants were administered a single test dose of RESP301 at the RTD of 4 mL. if tolerated and symptoms of exacerbation developed, eligible participants were to self-administer RESP301 TID for 7 days at the RTD.
Arm/Group | Part 0 | Part 1A - 1ml | Part 1A - 2ml | Part 1A - 3ml | Part 1A - 4ml | Part 1A - 5ml | Part 1A - 6ml | Part 1B - 6ml +SABA | Part 2 - RTD 4ml RTD 4ml RTD 4ml
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 1/8 | 4/16
Other Adverse Events (participants affected / at risk) | 4/4 | 4/8 | 4/8 | 1/8 | 5/8 | 5/8 | 4/6 | 6/8 | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 0 (N=4) | Part 1A - 1ml (N=8) | Part 1A - 2ml (N=8) | Part 1A - 3ml (N=8) | Part 1A - 4ml (N=8) | Part 1A - 5ml (N=8) | Part 1A - 6ml (N=6) | Part 1B - 6ml +SABA (N=8) | Part 2 - RTD 4ml RTD 4ml RTD 4ml (N=16)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
End stage COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lobar collapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compressed Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Severe Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 0 (N=4) | Part 1A - 1ml (N=8) | Part 1A - 2ml (N=8) | Part 1A - 3ml (N=8) | Part 1A - 4ml (N=8) | Part 1A - 5ml (N=8) | Part 1A - 6ml (N=6) | Part 1B - 6ml +SABA (N=8) | Part 2 - RTD 4ml RTD 4ml RTD 4ml (N=16)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 4 (5) | 1 (1) | 5 (5) | 5 (5) | 4 (4) | 6 (6) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT04858451/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04858451/SAP_001.pdf